CLINICAL TRIAL: NCT03318328
Title: Evaluation of Food Insecurity in Adults and Children With Cystic Fibrosis
Acronym: FI
Status: Completed | Type: Observational
Sponsor: Dixie Durham (Other)
Responsible Party: Sponsor-Investigator, Dixie Durham, Research Coordinator, St. Luke's Health System, Boise, Idaho
Organization: St. Luke's Health System, Boise, Idaho (Other)
Other Study IDs: 2017Food
Record Dates: First submitted 2017-10-16; First posted 2017-10-23 (Actual); Last update posted 2023-11-30 (Actual); Status verified 2023-11

CONDITIONS: Cystic Fibrosis
MeSH Terms: conditions — Cystic Fibrosis | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Other
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: survey

SUMMARY:
A survey of adults and parents of children with cystic fibrosis on food insecurity

DETAILED DESCRIPTION:
A survey of adults and parents of children with cystic fibrosis to determine any correlation between food insecurity and BMI or food insecurity and FEV1, and to determine what level of food insecurity is present.

ELIGIBILITY:
Inclusion Criteria: have CF and are willing to complete a questionnaire during a routine clinic visit

-

Exclusion Criteria:

* NA

Max Age: 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: adults and parents of children with cystic fibrosis
Sampling Method: Non-Probability Sample
Enrollment: 87 (Actual)
Dates: Start 2013-08-01 (Actual); Primary Completion 2015-03-31 (Actual); Study Completion 2015-03-31 (Actual)

PRIMARY OUTCOMES:
Evaluate food insecurity incidence in CF patients | one time questionnaire administered during a clinic visit
  Using a survey, determine the number of people who report food insecurity

SECONDARY OUTCOMES:
Determine if food insecurity leads to worse lung function in CF patients | one time questionnaire administered during a clinic visit
  Using a survey, report the current FEV1 and the number of people who report food insecurity to determine if there is a correlation
Determine if food insecurity leads to worse BMI in CF patients | one time questionnaire administered during a clinic visit.
  using a survey, report the current BMI and the number of people who report food insecurity to see if there is a correlation

IPD SHARING:
Plan to Share IPD: Undecided
undecided

REFERENCES:
- See also: Publication — https://www.frontiersin.org/articles/10.3389/fpubh.2018.00348/full